CLINICAL TRIAL: NCT01028209
Title: Evaluation of [18F] PBR06 and PET as a Marker of Inflammation in Subjects With Neurological Conditions
Acronym: PBR06
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Institute for Neurodegenerative Disorders (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PBR06 001
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Alzheimer Disease; Parkinson Disease; Multiple Sclerosis
MeSH Terms: conditions — Alzheimer Disease; Parkinson Disease; Multiple Sclerosis | interventions — N-fluoroacetyl-N-(2,5-dimethoxybenzyl)-2-phenoxyaniline

ARMS (1):
- Assess [18F] PBR06 and PET imaging (Experimental)
  Interventions: Drug: [18F] PBR06

INTERVENTIONS:
Drug: [18F] PBR06 — Subjects will be injected with 5mCi, not to exceed >10% of 5mCI, of [18F]PBR06, followed by PET imaging.

SUMMARY:
The underlying goal of this study is to assess [18F] PBR06 PET imaging as a tool to detect microglial activation in the brain of Alzheimer Disease (AD), Parkinson Disease (PD) and Multiple Sclerosis (MS) research participants.

ELIGIBILITY:
Inclusion Criteria:

* The following criteria will be met for inclusion of AD subjects in this study:

  * The participant is 50 years or older.
  * Written informed consent is obtained.
  * Participants have a clinical diagnosis of probable Alzheimer's disease based on National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) criteria.
  * Clinical Dementia Rating Scale score ≤ 2.
  * Modified Hachinski Ischemia Scale score of ≤ 4.
  * For females, non-child bearing potential or a negative urine or blood pregnancy test on day of [18F]-PBR06 injection.
* The following criteria will be met for inclusion of PD subjects in this study:

  * The participant is 30 years or older.
  * Written informed consent is obtained.
  * Participants have a clinical diagnosis of Parkinson disease (at least two of the three cardinal symptoms: resting tremor, rigidity, bradykinesia).
  * Hoehn and Yahr ≤4.
  * For females, non-child bearing potential or a negative urine or blood pregnancy test on day of [18F]-PBR06 injection.
* The following criteria will be met for inclusion of MS subjects in this study:

  * The participant is 18 years or older.
  * Written informed consent is obtained.
  * Participants have a clinical diagnosis of Multiple Sclerosis (per the 2005 Revised McDonald Criteria; Polman, et al., 2005).
  * Kurtzke Expanded Disability Status Scale (EDSS) ≤ 7.5.
  * For females, non-child bearing potential or a negative urine or blood pregnancy test on day of [18F]-PBR06 injection
* The following criteria will be met for inclusion of healthy control subjects in this study:

  * The participant is 18 years or older.
  * Written informed consent is obtained.
  * Negative history of neurological or psychiatric illness based on evaluation by a research physician.
  * Clinical Dementia Rating score = 0.
  * For females, non-child bearing potential a negative urine or blood pregnancy test on day of [18F]-PBR06 injection.

Exclusion Criteria:

* Alzheimer's subjects will be excluded from participation for the following reasons:

  * The subject has a history of significant cerebrovascular disease.
  * The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness
  * The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
  * Pregnancy
* Parkinson's subjects will be excluded from participation for the following reasons:

  * The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness
  * The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
  * Pregnancy
* MS subjects will be excluded from participation for the following reasons:

  * The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness
  * The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
  * Pregnancy
* Healthy control subjects will be excluded from participation for the following reasons:

  * The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness.
  * The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
  * Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-09-22 (Actual); Study Completion 2010-09-22 (Actual)

PRIMARY OUTCOMES:
To evaluate [18F] PBR06 PET imaging as a tool to detect microglial activation in the brain of AD, PD and MS research participants. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Danna Jennings, MD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (1):
- Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States